CLINICAL TRIAL: NCT02572687
Title: An Open-Label, Multicenter, Phase 1 Study of Ramucirumab Plus MEDI4736 in Patients With Locally Advanced and Unresectable or Metastatic Gastrointestinal or Thoracic Malignancies
Brief Title: A Study of Ramucirumab (LY3009806) Plus MEDI4736 in Participants With Advanced Gastrointestinal or Thoracic Malignancies
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Collaborators: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 16116; I4T-MC-JVDJ (Other: Eli Lilly and Company); 2015-003013-14 (EudraCT Number)
Record Dates: First submitted 2015-10-07; First posted 2015-10-09 (Estimated); Last update posted 2021-01-20 (Actual); Status verified 2021-01

CONDITIONS: Gastric Cancer; Gastroesophageal Junction Adenocarcinoma; Non-Small Cell Lung Cancer; Hepatocellular Carcinoma
Keywords: metastatic; advanced; immuno-oncology; vascular endothelial growth factor (VEGF); angiogenesis; PD-1; PD-L1
MeSH Terms: conditions — Stomach Neoplasms; Carcinoma, Non-Small-Cell Lung; Carcinoma, Hepatocellular; Neoplasm Metastasis | interventions — Ramucirumab; durvalumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Ramucirumab + MEDI4736 (NSCLC) (Experimental): In phase 1a (DLT phase), ramucirumab plus MEDI4736 given intravenously (IV) every 3 weeks (q3w) of a 21 day treatment cycle. Participants may continue to receive study treatment until discontinuation criteria are met.
  In phase 1b (expansion phase), ramucirumab plus MEDI4736 given IV q3w. Participants may continue to receive study treatment until discontinuation criteria are met.
  Interventions: Drug: Ramucirumab; Drug: MEDI4736
- Ramucirumab + MEDI4736 (Gastric/GEJ) (Experimental): In phase 1a (DLT phase), ramucirumab plus MEDI4736 given IV every 2 weeks (q2w) of a 28 day treatment cycle. Participants may continue to receive study treatment until discontinuation criteria are met.
  In phase 1b (expansion phase), ramucirumab plus MEDI4736 given IV q2w. Participants may continue to receive study treatment until discontinuation criteria are met.
  Interventions: Drug: Ramucirumab; Drug: MEDI4736
- Ramucirumab + MEDI4736 (HCC) (Experimental): In phase 1a (DLT phase), ramucirumab plus MEDI4736 given IV q2w of a 28 day treatment cycle. Participants may continue to receive study treatment until discontinuation criteria are met.
  In phase 1b (expansion phase), ramucirumab plus MEDI4736 given IV q2w. Participants may continue to receive study treatment until discontinuation criteria are met.
  Interventions: Drug: Ramucirumab; Drug: MEDI4736

INTERVENTIONS:
Drug: Ramucirumab — Administered IV
  Other Names: LY3009806; IMC-11121B; Cyramza
Drug: MEDI4736 — Administered IV

SUMMARY:
The main purpose of this study is to evaluate the safety of ramucirumab plus MEDI4736 in participants with locally advanced and unresectable or metastatic gastrointestinal or thoracic malignancies including gastric or gastroesophageal junction (GEJ) adenocarcinoma, non-small cell lung cancer (NSCLC), or hepatocellular carcinoma (HCC).

ELIGIBILITY:
Inclusion Criteria:

* Measurable metastatic disease or locally advanced and unresectable disease

  * Has histopathologically confirmed gastric or GEJ adenocarcinoma with documented disease progression after 1-2 prior lines of systemic therapy
  * Has histopathologically confirmed nonsquamous or squamous NSCLC with documented disease progression after 1-3 prior lines of systemic therapy
  * Has histopathologically or cytologically confirmed HCC, Child-Pugh Class A, with documented disease progression during or after discontinuation of sorafenib therapy, or intolerance of sorafenib therapy, and an α-fetoprotein (AFP) ≥ 1.5x upper limit of normal
* Availability of tumor tissue for biomarker analysis
* Has an Eastern Cooperative Oncology Group Performance Status of 0 or 1
* Has adequate organ function

Exclusion Criteria:

* Has known brain metastases
* Has a history of prior cancers not included in this study that were either not treated with curative intent or have been active within the past 5 years
* History of allogeneic organ transplant
* Has active or prior documented autoimmune disease within the past 24 months
* Has human immunodeficiency virus (HIV) infection or acquired immunodeficiency syndrome (AIDS)-related illness, or a history of immunodeficiency
* Has active hepatitis B or hepatitis C infection, or co-infection with both hepatitis B and C virus
* For gastric/GEJ and NSCLC participants, has chronic hepatitis B or hepatitis C infection. (For HCC participants, those with chronic hepatitis B virus [HBV] infection with a negative HBV deoxyribonucleic acid [DNA] test and who are on antiviral therapy, and those with chronic hepatitis C virus [HCV] infection are eligible)
* Has a history of interstitial lung disease, idiopathic pulmonary fibrosis, pneumoconiosis, non-infections pneumonitis, radiation-induced or drug-induced pneumonitis
* Has received any previous systemic therapy targeting programmed death (PD) 1 or PD-ligand 1/2 signaling pathways, and other immune checkpoint inhibitors
* Have received previous systemic therapy with ramucirumab

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 85 (Actual)
Dates: Start 2016-02-19 (Actual); Primary Completion 2018-03-27 (Actual); Study Completion 2021-01-13 (Actual)

PRIMARY OUTCOMES:
Number of Participants with Dose Limiting Toxicities (DLTs) | Cycle 1 (up to 28 days)

SECONDARY OUTCOMES:
Percentage of Participants with a Best Response of Complete Response (CR) or Partial Response (PR): Objective Response Rate (ORR) | Baseline to Disease Progression (Approximately 22 Months)
Proportion of Participants with a Best Overall Response of CR, PR, or Stable Disease (SD): Disease Control Rate (DCR) | Baseline to Disease Progression (Approximately 22 Months)
Duration of Response (DoR) | Date of CR or PR to Date of Objective Disease Progression or Death Due to Any Cause (Approximately 22 Months)
Time to First Response (TTR) | Baseline to Date of CR or PR (Approximately 22 Months)
Progression Free Survival (PFS) | Baseline to Progressive Disease or Death from Any Cause (Approximately 22 Months)
Overall Survival (OS) | Baseline to Progressive Disease or Death from Any Cause (Approximately 32 Months)
Pharmacokinetics (PK): Maximum Concentration (Cmax) of Ramucirumab and MEDI4736 | Predose Cycle 1 Day 1 through Follow Up (Approximately 22 Months)
PK: Minimum Concentration (Cmin) of Ramucirumab and MEDI4736 | Predose Cycle 1 Day 1 through Follow up (Approximately 22 Months)
Number of Participants with Treatment Emergent Anti Ramucirumab Antibodies | Predose Cycle 1 Day 1 through Follow Up (Approximately 22 Months)
Number of Participants with Treatment Emergent Anti MEDI4736 Antibodies | Predose Cycle 1 Day 1 through Follow Up (Approximately 22 Months)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (25):
- United States (7):
  - UCLA Medical Center, Santa Monica, California
  - Johns Hopkins University, Baltimore, Maryland
  - Washington University Medical Center, St Louis, Missouri
  - Carolinas Medical Center, Charlotte, North Carolina
  - The Miriam Hospital, Providence, Rhode Island
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - University of Texas MD Anderson Cancer Center, Houston, Texas
- France (4):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Besançon
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Marseille
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Montpellier
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Saint-Etienne
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Großhansdorf, Germany
- Israel (3):
  - Hadassah Medical Center - Ein Karem, Jerusalem
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Ramat Gan
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Tel Aviv
- Italy (2):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Milan
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Rozzano
- South Korea (2):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician, Seoul
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Seoul
- Spain (3):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Madrid
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Málaga
  - Hospital Virgen del Rocío, Seville
- Taiwan (3):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Tainan
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician, Tainan
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Taipei

REFERENCES:
- See also: A Study of Ramucirumab (LY3009806) Plus MEDI4736 in Participants With Advanced Gastrointestinal or Thoracic Malignancies — https://trials.lillytrialguide.com/en-US/trial/1MGivPlaAo26qYOuKOGOAe?conditionId=6BrOA7cZt6ESK8AScGGEao